CLINICAL TRIAL: NCT04835727
Title: Effect of Semi-vegetarian Diet in Inflammatory Bowel Disease Patients With Clinical Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Assistant Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Si 063/2020
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases; Calprotectin; Fecal Microbiota; Vegetarian Diet
Keywords: Vegetarian diet; inflammatory bowel diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective interventional cohort study in patients with clinically quiescent IBD. At enrollment, clinical information, dietary intake, inflammatory markers, and fecal microbiota were recorded. Dietary intake was assessed by an experienced nutritionist using pictures of food, a dietary questionnaire, and patient interviewing. The nutritionist advised the participants to intake a semi-vegetarian diet and increase dietary fiber consumption. The changes in clinical symptoms, dietary intake, inflammatory markers, and fecal microbiota were recorded in each visit for 1 year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-vegetarian diet (Experimental): All patients in this study will be advised by an experienced nutritionist to intake high fiber diets with a low intake of red meat and processed food.
  Interventions: Other: Semi-vegetarian diet and increase fiber consumption

INTERVENTIONS:
Other: Semi-vegetarian diet and increase fiber consumption — All patients in this study will be advised by an experienced nutritionist to intake high fiber diets with a low intake of red meat and processed food.

SUMMARY:
In the 21st century, the incidence of inflammatory bowel disease (IBD) globally increases. Higher incidence of IBD development may implicate that environmental factors played essential roles in IBD pathogenesis. One of the environmental factors is a westernized diet that contains a high amount of animal protein and a low amount of dietary fiber. This kind of diet can lead to gut microbial dysbiosis and increase susceptibility to IBD. A microbial dysbiosis pattern in IBD is a decrease in microbial diversity and the inversed ratio of local protective and pathologic bacteria. High animal protein was associated with an increased risk of IBD and increased risk of disease relapse meanwhile dietary fiber was associated with IBD risk reduction. A semi-vegetarian diet is a diet with high fiber and low red meat and processed food that may reduce inflammatory activity in IBD. The study in the semi-vegetarian diet in IBD activity is still limited.

This study aimed to evaluate a semi-vegetarian diet's effect in maintaining IBD remission in disease quiescence patients.

DETAILED DESCRIPTION:
This study is a prospective interventional cohort in clinically quiescence IBD patients in Siriraj Hospital, Mahidol University, Bangkok, Thailand. At enrollment, clinical information, dietary intake, inflammatory markers, and fecal microbiota will be recorded. Dietary intake will be assessed by an experienced nutritionist using pictures of food, a dietary questionnaire, and patient interviewing. The nutritionist advises the participants to consume a semi-vegetarian diet which includes high dietary fiber consumption and low red meat and processed food consumption. All patients will be required to send all pictures of food intake three days in 1 week before every visit, including two weekdays and one weekend. The dietary component will be analyzed using Nutrient calculation computer software INMUCAL-Nutrient V3 database NB1 (Institute of Nutrition, Mahidol University. Nakornpathom. 2013). The study will take 1 year including 6 visits (including baseline, 6th weeks, 18th week, 30th week, 42nd week, 54th week) for each patient. The primary outcome is the effect of increasing fiber diets and decreasing red meat and processed food on maintaining clinical remission in IBD. Secondary outcomes are the effect of modifying diet on change of inflammatory markers, microbiota, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Crohn's disease or Ulcerative colitis
2. Age ≥ 18 years old
3. Disease in remission at least 2weeks by following criteria Crohn's disease: Crohn's Disease Activity Index(CDAI) < 150 Ulcerative colitis: Mayo Ulcerative Colitis Subscore ≤ 2
4. Prednisolone ≤ 15 mg/day for at least 1 month
5. Stable immunomodulator dosage at least 1 month
6. Stable biologic agent at least 2 months

Exclusion Criteria:

1. Patients with Ulcerative colitis with a history of proctocolectomy
2. Patients with Crohn's disease with bowel stricture
3. Patients with recently antibiotic usage within 1 month
4. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of participants with clinical relapses | 1 year
  Effect of semi-vegetarian food consumption on the rate of participants with clinical relapses assessed by Crohn's disease activity index for Crohn's disease and the clinical Mayo Score or partial Mayo Score for ulcerative colitis. The Crohn's disease activity index ranges from 0 to 1100, a higher score means a worse outcome, and clinical relapse is defined if the score is at least 150 points. The clinical Mayo Score for ulcerative colitis ranges from 0 to 9, a higher score means a worse outcome, and clinical relapse is defined if the score is at least 2 points.

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) | 1 year
  Effect of semi-vegetarian food consumption on inflammatory markers levels including serum CRP
fecal calprotectin level | 1 year
  Effect of semi-vegetarian food consumption on inflammatory markers levels including fecal calprotectin level
Fecal microbiota | 1 year
  Effect of semi-vegetarian food consumption on changing of fecal microbiota composition and diversity (Shannon's diversity index)
Quality of life score of SIBDQ | 1 year
  Effect of semi-vegetarian food consumption on quality of life: SIBDQ
Quality of life score of EQ5D3L | 1 year
  Effect of semi-vegetarian food consumption on quality of life: EQ5D3L

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand